CLINICAL TRIAL: NCT00351247
Title: Clinical and MRI Evaluation of 2 Vs 4 Cycles of Postconditioning During Primary PCI With Direct Stenting
Brief Title: Postconditioning in Primary PCI and Direct Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4066-VG-CTIL
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-07

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Primary PCI; Postconditioning; MRI
MeSH Terms: conditions — Myocardial Infarction | interventions — Ischemic Postconditioning

INTERVENTIONS:
Procedure: Postconditioning

SUMMARY:
To determine the safety and efficacy of 2 vs 4 cycles of postconditioning method during primary PCI and direct stenting in acute MI, and to compared to primary PCI and direct stenting without the postconditioning.

DETAILED DESCRIPTION:
Sample size: 45 subjects

Site Locations: Sheba medical center

Patients: Patients presenting with an acute MI with onset of symptoms  6h, and planned to undergo primary PCI will be included. The target lesion should be located in the proximal or middle segment of a main native coronary artery, and should be suitable for percutaneous intervention.

Primary Objective: To determine the safety and efficacy of 2 vs 4 cycles of postconditioning method during primary PCI and direct stenting in acute MI, and to compared to primary PCI and direct stenting without the postconditioning.

Primary Endpoint:

* ST segment resolution.
* Segmental wall motion score, resolution of edema and wall thickness by echocardiography.
* Infarct size estimation by cardiac enzymes and cardiac MRI.

Secondary endpoints:

* Composite endpoint of Major Adverse Cardiac Events (MACE) at 30 and 90 days

Methods:

* ECG at baseline, immediately after procedure, 90 and 180 minutes after the procedure and 6-24 hours after intervention.
* Core laboratory angiography measurements of TIMI flow, corrected TIMI Frame count, myocardial blush score and left ventricular angiography.
* Myocardial enzymes measurements: every 4 hours in the first 24 hours and every 6 hours in the following 48 hours.
* Left ventricular ejection fraction and wall motion score determined by echocardiography.
* Cardiac MRI estimation of infarct size. • Clinical follow-up at 30 and 90 days post procedure.

Follow-up:

* Follow up at 30 days: Clinical.
* Clinical Follow up & Cardiac MRI at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 21 years of age and provides informed consent.
* Evidence of AMI as indicated by signs and symptoms. Diagnosis of ST-segment elevation AMI will be based on chest pain for >30 minutes and ST-segment elevation of >1mV in 2 limb lead or >2mV in 2 anterior leads contiguous leads on the 12-lead ECG.
* Eligible to undergo primary PCI.
* Symptom duration is < 6 hours prior to primary PCI.
* Angiographic: The target lesion in the infarct related artery (IRA) should be occluded (TIMI).
* Angiographic: The target lesion in the proximal or middle segment of a native major coronary artery (LAD, RCA or dominant CX).
* Angiographic: The target lesion should be suitable for PTCA or stenting.
* Angiographic: The IRA occlusion will be successfully opened by stenting with TIMI 2-3

Exclusion Criteria:

* Unwillingness to participate.
* Prior Acute MI
* Cardiac arrest or Killip score III-IV
* Women with known pregnancy.
* Active significant bleeding.
* Known allergy for aspirin, ticlopidine and clopidogrel, or heparin.
* Chronic renal failure with creatinine > 2 mg/dl
* Other medical illness associated with limited life expectancy or that may cause the patient to be non-compliant with the protocol.
* Current participation in other trials using investigational drugs or devices.
* Contraindications to MRI including: arrythmias, cardiac pacer, brain aneurysm clips, cochlear implants, nerve stimulator.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2006-07; Study Completion 2007-05

PRIMARY OUTCOMES:
ST segment resolution.
Segmental wall motion score, resolution of edema and wall thickness by echocardiography.
Infarct size estimation by cardiac enzymes and cardiac MRI.

SECONDARY OUTCOMES:
Composite endpoint of Major Adverse Cardiac Events (MACE) at 30 and 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Victor Guetta, MD, Principal Investigator — Sheba Medical Center; Jonathan Leor, MD, Principal Investigator — Neufeld Cardiac Research Center; Elad Maor, MD, Principal Investigator — Neufeld Cardiac Research Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Staat P, Rioufol G, Piot C, Cottin Y, Cung TT, L'Huillier I, Aupetit JF, Bonnefoy E, Finet G, Andre-Fouet X, Ovize M. Postconditioning the human heart. Circulation. 2005 Oct 4;112(14):2143-8. doi: 10.1161/CIRCULATIONAHA.105.558122. Epub 2005 Sep 26. PMID 16186417
- [Background] Zhao ZQ, Corvera JS, Halkos ME, Kerendi F, Wang NP, Guyton RA, Vinten-Johansen J. Inhibition of myocardial injury by ischemic postconditioning during reperfusion: comparison with ischemic preconditioning. Am J Physiol Heart Circ Physiol. 2003 Aug;285(2):H579-88. doi: 10.1152/ajpheart.01064.2002. PMID 12860564